CLINICAL TRIAL: NCT03202563
Title: A Multicenter, Randomized, Active-controlled, Parallel Group, Open-label, Phase 4 Trial to Evaluate the Efficacy on Glycemic Variability and Safety of Gemigliptin 50mg q.d., Versus Dapagliflozin 10mg q.d. Added to Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Alone or Diabetes Medication Naïve Patient
Brief Title: Trial to Evaluate the Efficacy on Glycemic Variability and Safety of Gemigliptin Compared With Dapagliflozin Added on Metformin Alone or Diabetes Medication Naïve Patient in Type 2 Diabetes Mellitus (Stable II Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL017
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444; dapagliflozin; Continuous Glucose Monitoring; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemigliptin 50mg (Experimental): the subjects should visit a study site 4 times during the treatment period for about 12 weeks in total.
  Drug: Gemigliptin Drug: Metformin Procedure: Diet/exercise questionnaire Procedure: Continuous Glucose Monitoring System(CGMS)
  Interventions: Drug: Gemigliptin 50mg; Procedure: Diet/exercise questionnaire; Device: Continuous Glucose Monitoring System(CGMS); Drug: Metformin
- Dapagliflozin 10mg (Active Comparator): the subjects should visit a study site 4 times during the treatment period for about 12 weeks in total.
  Drug: Dapagliflozin Drug: Metformin Procedure: Diet/exercise questionnaire Procedure: Continuous Glucose Monitoring System(CGMS)
  Interventions: Drug: Dapagliflozin 10mg; Procedure: Diet/exercise questionnaire; Device: Continuous Glucose Monitoring System(CGMS); Drug: Metformin

INTERVENTIONS:
Drug: Gemigliptin 50mg — For patients who have been randomized to Gemigliptin(Experimental arm), the patients continue to take a gemigliptin 50mg 1 tablet by once daily during study treatment period(Visit 3(day 1)~Visit 6(day 91))
  Arms: Gemigliptin 50mg
Drug: Dapagliflozin 10mg — For patients who have been randomized to Dapagliflozin(Active Comparator arm), the patients continue to take a dapagliflozin 10mg 1 tablet by once daily during study treatment period(Visit 3(day 1)~Visit 6(day 91))
  Arms: Dapagliflozin 10mg
Procedure: Diet/exercise questionnaire — doing exercise with about intermediate intensity(50~70%) for ≥150minutes in total over at least 3 times(every other day) weekly should be recommended and regular diet without greater changes in life style as much as possible during the whole study period.
  the questionnaire regarding diet/exercise will be collected at -day 6, day 1, day29, day85, day 91
Device: Continuous Glucose Monitoring System(CGMS) — For patients who have been screening completely, the subjects will be attached CGMS(ipro-2) twice from Visit 2(-day 6) to Visit 3(day 1) and Visit 5(day 85) to Visit 6(day 91)
Drug: Metformin — For patients who have been taking metformin, the patients who had taken at least 1000 mg of metformin daily and continue the same dosage and administration as before participant in the study

SUMMARY:
The objective of this study is to evaluate the efficacy on glycemic variability and safety of gemigliptin 50 mg orally administered once daily for 12 weeks compared with Dapagliflozin 10mg in patients with type 2 diabetes mellitus who have inadequate glycemic control on metformin alone or diabetes medication naïve patient

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus of 20~70years of age at the time of Visit 1 (Screening)
2. Patients with HbA1c measured in the local lab ranged from 7 to 11%satisfying the following conditions at the time of Visit 1(Screening)

   * Type 2 diabetes mellitus medication naïve patients or patients who had not taken diabetes medication other than metformin within 8 weeks prior to Visit 1(Screening)
   * For patients who have been taking metformin alone within 12 weeks prior to visit 1(Screening) and had taken at least 1000 mg of metformin daily without dose adjustment for 4 weeks prior to Visit 1(Screening)
3. Patients who have signed an informed consent themselves after receiving explanation about the objectives, methods, effects, etc. of the clinical study
4. Patients who are applicable to one of the three in the following. 1) Surgically infertile patients 2) Postmenopausal female patients of ≥45 years of age for whom ≥2 years elapsed since their last menstruation 3) Premenopausal fertile female patients or surgically non-infertile male patients who have agreed to use at least 2 kinds of contraceptive measures (certainly including one of the barrier methods) to avoid pregnancy until 14 days after the last dose of the investigational product

   * Barrier methods: Condom, Diaphragm, Cervical cap(Pessary), Spermicide
   * Hormonal methods: Pills, Injection(Depot), Skin patch, Hormonal implant(Implanon), Vaginal ring
   * Intrauterine Devices(IUDs): Cooper IUD(Loop), Hormonal IUD(Mirena)
   * Natural methods: Basic body temperature, Ovulation period, Coitus interruptus, Abstinence

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus*, Diabetic ketoacidosis, Diabetic coma, Diabetic pre-coma
2. Patients with Gestational diabetes, or secondary diabetes
3. Patients with Body Mass Index(BMI) >40 kg/m2 at the time of Visit 1(Screening)
4. Patients with a history of the following

   * Patients with NYHA Class III, IV congestive heart failure or arrhythmia requiring treatment at the time of Visit 1(Screening)
   * Patients whose TSH level is out of the normal range and who have thyroidal dysfunction requiring drug therapy at the time of Visit 1(Screening) (However, those who have been taking thyroid hormone at a fixed dose since previous 6 weeks prior to Visit 1[Screening] and whose TSH level is within the normal range can participate in the study.)
   * Patients with a glomerular filtration rate (eGFR) less than 60 mL/min /1.73 m2, dnd stage renal disease, dialysis or with renal disease that may result from conditions such as cardiovascular shock, acute myocardial infarction and sepsis, or patients with renal insufficiency at the time of Visit 1(Screening)
   * Patients who are receiving intravenous iodine contrast agents at the time of visit 1(Screening) or planned during the clinical trial period (eg, intravenous urography, venous cholangiography, angiography, computed tomography using contrast media, etc.) ). For patients who have received this test, they can re-evaluate the renal function 48 hours after the test and only participate in clinical trials after they have been found to be normal.
   * Patients with pulmonary embolism, severe pulmonary dysfunction, or who are susceptible to be accompanied by hypoxemia at the time of Visit 1(Screening)
   * Patients on drug therapy due to gastrointestinal disturbance including dehydration, diarrhea, and vomiting at the time of Visit 1(Screening) Patients with severe infection or severe trauma at the time of Visit 1(Screening)
   * Patients with malnutrition status, starvation status, weakness status, pituitary insufficiency or adrenal insufficiency at the time of Visit 1(Screening)
   * Patients with a history of diabetic ketoacidosis or hyperosmolar non-ketotic coma within 12 weeks prior to Visit 1(Screening)
   * Patients with a history of myocardial infarction, unstable angina, and coronary artery bypass graft(CABG) within 12 weeks prior to Visit 1(Screening)
   * Patients who had had a surgical operation within 4 weeks prior to Visit 1(Screening) (excluding minor surgeries without restriction on food and fluid intake) or who are scheduled to have a significant surgery during the study period
   * Patients with a history of alcoholism or drug addiction within 12weaks prior to Visit 1(Screening)
   * Patients with a history of malignant tumors within 5 years prior to Visit 1(Screening). However, patients with basal cell or squamous cell skin cancer, or in situ cervical cancer treated properly can participate in the study.
5. Patients with the outcomes of the laboratory tests performed at Visit 1(Screening) applicable to the criteria below

   * Bilirubin >2 × upper limit of normal(ULN)
   * AST/ALT >3 × ULN
6. Patients with a history of hypersensitivity reactions to the drugs below

   * Gemigliptin or drugs belonging to dipeptidyl-peptidase4(DPP4) inhibitors
   * Dapagliflozin or drugs belonging to Sodium/glucose co transport-2(SGLT-2) inhibitor
   * Metformin or drugs belonging to biguanides
7. Patients who were administered the drugs below

   * Patients who had been administered anti-obesity drugs within 4 weeks prior to Visit 1(Screening)
   * Patients who had been administered insulin or GLP-1 analogues within 8 weeks prior to Visit 1(Screening)
   * Patients who had been administered warfarin, dicoumarin, and digoxin within 4 weeks prior to Visit 1(Screening)
   * Patients who are being administered any of the strong CYP3A4 inducers (rifampicin[rifampin], dexamethasone, phenytoin, carbamazepine, rifabutin, phenobarbital) at the time of Visit 1(Screening)
   * Patients who had been being administered glucocorticoids continuously within 2 weeks prior to Visit 1(Screening) or who are required to take glucocorticoids continuously in the future
8. Patients with a genetic problems such as Galactose intolerance, Lapp lactose deficiency, Glucose-galactose malabsorption)
9. Female patients who are pregnant or lactating
10. Patients who have an experience of participation in another clinical study within 12 weeks prior to Visit1(screening)
11. Patients who are otherwise considered to be ineligible for this study on investigators' judgment

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline MAGE(Mean amplitude of glycemic excursion) at week 12 | baseline (visit 2~visit3) and week 12 (visit 5~visit 6)
  MAGE will be calculated from MBG which has been measured by CGMS(Continuous Glucose Monitoring System) during CGM period(visit 2~visit 3, visit 5~visit 6)

SECONDARY OUTCOMES:
Changes from baseline MBG(Mean Blood Glucose) at week 12 | baseline (visit 2~visit3) and week 12 (visit 5~visit 6)
  MBG is a mean blood glucose measured by CGMS(Continuous Glucose Monitoring System) during CGM period(visit 2~visit 3, visit 5~visit 6)
Changes from baseline SD(Standard Deviation) at week 12 | baseline (visit 2~visit3) and week 12 (visit 5~visit 6)
  SD is a standard deviation of MBG measured by CGMS(Continuous Glucose Monitoring System) during CGM period(visit 2~visit 3, visit 5~visit 6)
Changes from baseline CV(Coefficient of variance) at week 12 | baseline (visit 2~visit3) and week 12 (visit 5~visit 6)
  CV is a coefficient of variance which is MBG divided by SD measured by MBG during CGM period(visit 2~visit 3, visit 5~visit 6)
Changes from baseline hsCRP at week 12 | baseline (visit 2) and week 12 (visit 5)
Changes from baseline Nitrotyrosine at week 12 | baseline (visit 2) and week 12 (visit 5)

OTHER OUTCOMES:
Changes of HbA1c at each visit | baseline(visit 2), week 5(visit 4), week 13(visit 5)
  values of parameters at the corresponding visit - values of parameters at visit 2(baseline)
Changes of Fasting plasma glucose at each visit | baseline(visit 2), week 5(visit 4), week 13(visit 5)
  values of parameters at the corresponding visit - values of parameters at visit 2(baseline)
Changes of Fasting serum insulin at each visit | baseline(visit 2), week 5(visit 4), week 13(visit 5)
  values of parameters at the corresponding visit - values of parameters at visit 2(baseline)
Changes of Glycated albumine at each visit | baseline(visit 2), week 5(visit 4), week 13(visit 5)
  values of parameters at the corresponding visit - values of parameters at visit 2(baseline)
Changes of baseline HOMA-β at week 13 | baseline(visit 2), week 13(visit 5)
Changes of baseline HOMA-IR at week 13 | baseline(visit 2), week 13(visit 5)
Changes of baseline LDL-C at week 13 | baseline(visit 2), week 13(visit 5)
Changes of baseline HDL-C at week 13 | baseline(visit 2), week 13(visit 5)
Changes of baseline Total Cholesterol at week 13 | baseline(visit 2), week 13(visit 5)
Changes of baselineTriglyceride at week 13 | baseline(visit 2), week 13(visit 5)
Changes of baseline BMI at week 13 | baseline(visit 2), week 13(visit 5)
Changes of baseline Body weight at week 13 | baseline(visit 2), week 13(visit 5)

CONTACTS AND LOCATIONS:
Overall Officials: Jaehyen Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided